CLINICAL TRIAL: NCT01426880
Title: A Randomized Phase II Trial Investigating the Addition of Carboplatin to Neoadjuvant Therapy for Triple-negative and HER2-positive Early Breast Cancer
Brief Title: Addition of Carboplatin to Neoadjuvant Therapy for Triple-negative and HER2-positive Early Breast Cancer
Acronym: GeparSixto
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: Teva Pharmaceuticals USA (Industry); Roche Pharma AG (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBG 66; 2011-000553-23 (EudraCT Number)
Record Dates: First submitted 2011-08-17; First posted 2011-09-01 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Tubular Breast Cancer Stage II; Mucinous Breast Cancer Stage II; Breast Cancer Female NOS; Invasive Ductal Breast Cancer; Tubular Breast Cancer Stage III; HER-2 Positive Breast Cancer; Inflammatory Breast Cancer Stage IV; Inflammatory Breast Cancer
Keywords: GBG; German Breast Group; neo-adjuvant; GBG Forschungs GmbH; Tubular breast cancer stage II; Mucinous breast cancer stage II; Invasive ductal breast cancer; Tubular breast cancer stage III; HER-2 positive breast cancer; Inflammatory breast cancer stage IV; Inflammatory breast cancer
MeSH Terms: conditions — Carcinoma, Ductal, Breast; Inflammatory Breast Neoplasms | interventions — Carboplatin; Bevacizumab; Paclitaxel; Doxorubicin; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carboplatin + background treatment (Experimental): Carboplatin AUC 2 min/mL weekly, infusion will be used as Add-on to the background therapy (same as comparator arm)
  Interventions: Drug: Carboplatin; Drug: background treatment
- background treatment only (Active Comparator): background treatment with NLPD (Myocet), Paclitaxel, Herceptin (Trastuzumab fpr Her2 pos), Tyverb (Lapatinib for Her2 pos), Avastin (Bevacizumab for triple negative) agents are used according to marketed formulation via normal procedures at each site and applied according to recommendations of the manufacturers.
  Interventions: Drug: background treatment

INTERVENTIONS:
Drug: Carboplatin — Carboplatin, AUC, 2 min/mL weekly, infusion
  Other Names: platin
  Arms: Carboplatin + background treatment
Drug: background treatment — background treatment according to standards fpr triple negative and Her2pos breast cancer patients Paclitaxel: 80 mg/m² i.v. given weekly on day 1 q day 8 for 18 weeks. NPLD (Myocet®): 20 mg/m² weekly on day 1 q day 8 for 18 weeks Trastuzumab (only for HER2-positive patients): Loading dose: 8 mg/kg, Maintenance dose: 6 mg/kg, day 1 q day 22 for 6 cycles. Post-surgery: up to a total duration of 1 year according to current AGO guidelines Lapatinib 750 mg/day p.o. continuously for 18 weeks; in case of good tolerability (no CTC grade II toxicity except alopecia and nausea/vomiting) during the first cycle the dose may be escalated to 1000 mg.
  Bevacizumab: 15 mg/kg i.v., day 1 q day 22 for 6 cycles (only in TNBC patients).
  Other Names: Avastin; Paclitaxel; Myocet; Lapatinib; Bevacizumab

SUMMARY:
Study participants with primary breast cancer will receive a standard chemotherapy with an anthracycline and a taxane as well as trastuzumab in case of HER2-positive tumors at doses and duration in concordance to current treatment guidelines. Patients will be receive and benefit in addition currently not in the neoadjuvant setting registered medication as lapatinib or bevacizumab of which significant increases of cure (pCR) rates have been reported in previous phase III studies. Patients randomized to carboplatin will receive in addition to the described backbone therapies a potentially active agent which suggested synergy of efficacy with chemotherapies as well as targeted agents. Patients might have the risk of an increase in toxicities due to the added agents and will have additional burden due to investigations required for study participation. However, due to the severity of the underlying disease and the high risk of relapse and death due to the stage of disease, this increase in toxicity and burden appears less relevant compared to the potential higher efficacy and finally cure rate by the incorporated treatments.

DETAILED DESCRIPTION:
Anthracycline/taxane based combination chemotherapy of at least 18 weeks represents the standard of care in the neoadjuvant setting. In HER2-positive disease trastuzumab is given simultaneously to chemotherapy. Recent data from the Neo-Altto and Neosphere trials suggest that a dual blockage of the HER2 receptor with e.g. trastuzumab and lapatinib reach significantly higher pCR rates than trastuzumab alone and should therefore represent the treatment back-bone of new neoadjuvant trials. A preplanned subgroup analysis of the GeparQuinto study demonstrated that in TNBC the addition of bevacizumab resulted in a significant increase of pCR rates (HR 1.4).

Having a better cardiac tolerability profile compared to conventional anthracyclines, the non-pegylated liposomal encapsulated doxorubicin (NPLD) Myocet® might provide the possibility to combine taxane, anthracycline, platinum salt as well with targeted agents as double HER2 blockage or bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* 1.Written informed consent for all study procedures according to local regulatory requirements prior to beginning specific protocol procedures.
* 2.Complete baseline documentation must be submitted via Medcodes® and approved by GBG Forschungs GmbH.
* 3.Unilateral or bilateral primary carcinoma of the breast, confirmed histologically by core biopsy. Fine-needle aspiration is not sufficient. Incisional biopsy is not allowed. In case of bilateral cancer, the investigator has to decide prospectively which side will be evaluated for the primary endpoint.
* 4.Tumor lesion in the breast with a palpable size of ≥ 2 cm or a sonographical size of ≥ 1 cm in maximum diameter. The lesion has to be measurable in two dimensions, preferably by sonography. In case of inflammatory disease, the extent of inflammation can be used as measurable lesion.
* 5.Patients should be in the following stages of disease: cT2 - cT4a-d or cT1c and cN+ or pNSLN+
* 6.In patients with multifocal or multicentric breast cancer, the largest lesion should be measured.
* 7.Centrally confirmed ER/PR/HER-2 and Ki-67 status detected on core biopsy. ER/PR positive is defined as >1% stained cells and HER2-positive is defined as HercepTest IHC 3+ or FISH ratio ≥ 2.2. Formalin-fixed, paraffin-embedded (FFPE) breast tissue from core biopsy has therefore to be sent to the Dept. of Pathology at the Charité, Berlin prior to randomization.
* 8.Age ≥ 18 years.
* 9.Karnofsky Performance status index ≥ 80%.
* 10.Normal cardiac function must be confirmed by ECG and cardiac ultrasound (LVEF or shortening fraction) within 3 months prior to randomization. LVEF must be above 55%.
* 11.Laboratory requirements: Hematology
* Absolute neutrophil count (ANC) ≥ 2.0 x 109 / L and
* Platelets ≥ 100 x 109 / L and
* Hemoglobin ≥ 10 g/dL (≥ 6.2 mmol/L) Hepatic function
* Total bilirubin < 1.5x UNL and
* ASAT (SGOT) and ALAT (SGPT) ≤ 1.5x UNL and
* Alkaline phosphatase ≤ 2.5x UNL. Renal function
* Creatinine ≤ 175 µmol/L (2 mg/dL) < 1.5x UNL
* Proteinuria: Urine dipstick for proteinuria < 2+. Patients discovered to have ≥ 2+ proteinuria on dipstick urinalysis should undergo a 24-hour urine collection and must demonstrate ≤ 1 g of protein in 24 hours. If creatinine is between 140 - 175 umol/L (1.6-2.0 mg/dL), the creatinine clearance (calculated or measured) should be ≥ 45 mL/min.
* 12.Negative pregnancy test (urine or serum) within 14 days prior to randomization for all women of childbearing potential.
* 13.Complete staging work-up within 3 months prior to randomization. All patients must have bilateral mammography, breast ultrasound (≤ 21 days), breast MRI (optional), chest X-ray (PA and lateral), abdominal ultrasound or CT scan or MRI, and bone scan done. In case of positive bone scan, bone X-ray (or CT or MRI) is mandatory. Other tests may be performed as clinically indicated.
* 14.Patients must be available and compliant for central diagnostics, treatment and follow-up.

Exclusion Criteria:

1. Prior chemotherapy for any malignancy.
2. Prior radiation therapy for breast cancer.
3. Pregnant or lactating patients. Patients of childbearing potential must implement adequate non-hormonal contraceptive measures (barrier methods, intrauterine contraceptive devices, sterilization) during study treatment.
4. Inadequate general condition (not fit for anthracycline-taxane-targeted agents-based chemotherapy).
5. Previous malignant disease being disease-free for less than 5 years (except CIS of the cervix and non-melanomatous skin cancer).
6. Known or suspected congestive heart failure (>NYHA I) and / or coronary heart disease, angina pectoris requiring antianginal medication, previous history of myocardial infarction, evidence of transmural infarction on ECG, uncontrolled or poorly controlled arterial hypertension (i.e. BP >160 / 90 mm Hg under treatment with two antihypertensive drugs), rhythm abnormalities requiring permanent treatment, clinically significant valvular heart disease.
7. Previous thromboembolic event (except when thrombophily screening is negative).
8. Known hemorrhagic diathesis or coagulopathy with increased bleeding risk.
9. History of significant neurological or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent
10. Pre-existing motor or sensory neuropathy of a severity ≥ grade 2 by NCI-CTC criteria v 4.0.
11. Currently active infection.
12. Active peptic ulcer.
13. Incomplete wound healing or unhealed bone fracture.
14. Disease significantly affecting gastrointestinal function, e.g. malabsorption syndrome, resection of the stomach or small bowel, ulcerative colitis.
15. History of abdominal fistula or any grade 4 non-gastrointestinal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months of enrolment.
16. Severe pulmonary condition / illness.
17. Major surgery within the last 28 days or anticipation of the need for major surgery during study treatment with bevacizumab. Minor surgeries including insertion of an indwelling catheter or sentinel lymph node biopsy within 24 h prior to chemotherapy.
18. Definite contraindications for the use of corticosteroids except inhalative corticoids.
19. Known hypersensitivity reaction to one of the compounds or incorporated substances used in this protocol;
20. Concurrent treatment with:

    * chronic corticosteroids unless initiated > 6 months prior to study entry and at low dose (≤ 10 mg methylprednisolone or equivalent).
    * sex hormones. Prior treatment must be stopped before study entry.
    * virostatic agents like sorivudine or analogs like brivudine, concurrent treatment with aminoglycosides.
    * anticoagulants: heparin, warfarin as well as acetylic acid (e.g. Aspirin®) at a dose of > 325 mg/day or clopidogrel at a dose of > 75 mg/day.
    * other experimental drugs or any other anti-cancer therapy.
    * drugs recognized as being strong inhibitors or inducers of the isoenzyme CYP3A, e.g. Rifabutin, Rifampicin, Clarithromycin, Ketoconazole, Itraconazole, Ritonavir, Telithromycin, Erythromycin, Verapamil, Diltiazem within the last 5 days or the expected need for these treatments during study participation.
21. Participation in another clinical trial with any investigational, not marketed drug within 30 days prior to study entry.
22. Male patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 2011-08; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Pathological complete response of breast and lymph nodes (ypT0 ypN0; primary endpoint) | 24 weeks (time window -3 weeks)
  Pathological response will be assessed considering all removed breast and lymphatic tissues from all surgeries. Surgery takes place shortly after the 18 weeks (six 3-week cycles) chemotherapy treatment. No microscopic evidence of residual viable tumor cells in all resected specimens of the breast and axilla meets the primary endpoint.

SECONDARY OUTCOMES:
1.ypT0/is ypN0; ypT0; ypT0/is; ypN0, and regression grades | 24 weeks (time window -3 weeks)
Clinical and imaging response | 24 weeks (time window -3 weeks)
  To determine the response rates of the breast tumor and axillary nodes based on physical examination and imaging tests. (sonography, mammography, or MRI) after treatment in both arms.
loco-regional invasive recurrence free survival (LRRFS), regional recurrence free survival (RRFS), local recurrence free survival (LRFS), distant-disease- free survival (DDFS), invasive disease-free survival (IDFS), and overall survival (OS) | 5 years
  LRRFS, RRFS, LRFS, DDFS, IDFS and OS are defined as the time period between registration and first event and will be analyzed after the end of the study by referring to data from GBG patient's registry.
Tolerability and Safety | during treatment 18 weeks
  Tolerability and Safety: Descriptive statistics for the 4 treatments will be given on the number of patients whose treatment had to be reduced, delayed or permanently stopped
pCR rates per arm | 24 weeks (time window -3 weeks)
  • To assess the pCR rates per arm separately in patients with triple-negative tumors and HER2-positive tumors.
Breast and axilla conservation rate | 24 weeks (time window -3 weeks)
  To determine the breast and axilla conservation rate after each treatment.
pCR rate and local recurrence free survival in correlation to clinical complete response and negative core biopsy before surgery | 5 years
  To determine the pCR rate and local recurrence free survival (LRFS) in patients with a clinical complete response (cCR) and a negative core biopsy before surgery.
Clinical and imaging response | 6 weeks
  To determine the response rates of the breast tumor and axillary nodes based on physical examination and imaging tests. (sonography, mammography, or MRI) after treatment in both arms.
PCR rate in patients with a clinical complete response and a negative core biopsy | 24 weeks (time window -3 weeks)
  To assess the pCR rate in patients with a clinical complete response and a negative core biopsy before surgery.
Regional recurrence free survival (RRFS)in patients with initial node-positive axilla | until event occurs - no events for cured patients
  To assess regional recurrence free survival (RRFS) in patients with initial node-positive axilla converted to negative at surgery and treated with sentinel node biopsy alone.
Examination and comparison of molecular markers | Baseline, 6 weeks and 24 weeks
  To examine and compare pre-specified molecular markers such as BRCA1-mRNA, P53, ALDH1, p4E-BP1, IL-8 metagene, B-Cell metagene as well as exploratory analyses and lymphocyte infiltration on core biopsies before and surgical tissue after end of chemotherapy. The aim is to identify potential predictive short and long term parameters.
CTC Substudy | Baseline, 6 weeks and 24 weeks
  To assess, characterize, and correlate circulating tumor cells and proteins with the effect of treatment.
Pharmacogenetic substudy | Baseline
  To correlate Single Nucleotide Polymorphisms (SNPs) of genes with the associated toxicity and histologically assessed treatment effect.
Ovarian Substudy | Baseline, 6 months, 12 months, 18 months, 24 months, 30 months
  To assess ovarian function measured by amenorrhea rate in correlation with changes in E2, FSH, Anti-Müller Hormone, ultrasound-follicle count in patients aged <45 years.

CONTACTS AND LOCATIONS:
Overall Officials: Gunter von Minckwitz, MD, Prof, Principal Investigator — ASCO, AACR, ESMO, DKG, DGGG, AGO, DGS, BIG, BCIRG, St. Gallen Consensus Panel
Locations (3):
- Germany (3):
  - Praxis Dr. Heinrich, Fürstenwalde, Brandenburg
  - Luisenkrankenhaus, Düsseldorf, North Rhine-Westphalia
  - NCT Heidelberg, Heidelberg

REFERENCES:
- [Result] Denkert C, von Minckwitz G, Brase JC, Sinn BV, Gade S, Kronenwett R, Pfitzner BM, Salat C, Loi S, Schmitt WD, Schem C, Fisch K, Darb-Esfahani S, Mehta K, Sotiriou C, Wienert S, Klare P, Andre F, Klauschen F, Blohmer JU, Krappmann K, Schmidt M, Tesch H, Kummel S, Sinn P, Jackisch C, Dietel M, Reimer T, Untch M, Loibl S. Tumor-infiltrating lymphocytes and response to neoadjuvant chemotherapy with or without carboplatin in human epidermal growth factor receptor 2-positive and triple-negative primary breast cancers. J Clin Oncol. 2015 Mar 20;33(9):983-91. doi: 10.1200/JCO.2014.58.1967. Epub 2014 Dec 22. PMID 25534375
- [Result] Loibl S, von Minckwitz G, Schneeweiss A, Paepke S, Lehmann A, Rezai M, Zahm DM, Sinn P, Khandan F, Eidtmann H, Dohnal K, Heinrichs C, Huober J, Pfitzner B, Fasching PA, Andre F, Lindner JL, Sotiriou C, Dykgers A, Guo S, Gade S, Nekljudova V, Loi S, Untch M, Denkert C. PIK3CA mutations are associated with lower rates of pathologic complete response to anti-human epidermal growth factor receptor 2 (her2) therapy in primary HER2-overexpressing breast cancer. J Clin Oncol. 2014 Oct 10;32(29):3212-20. doi: 10.1200/JCO.2014.55.7876. Epub 2014 Sep 8. PMID 25199759
- [Result] von Minckwitz G, Schneeweiss A, Loibl S, Salat C, Denkert C, Rezai M, Blohmer JU, Jackisch C, Paepke S, Gerber B, Zahm DM, Kummel S, Eidtmann H, Klare P, Huober J, Costa S, Tesch H, Hanusch C, Hilfrich J, Khandan F, Fasching PA, Sinn BV, Engels K, Mehta K, Nekljudova V, Untch M. Neoadjuvant carboplatin in patients with triple-negative and HER2-positive early breast cancer (GeparSixto; GBG 66): a randomised phase 2 trial. Lancet Oncol. 2014 Jun;15(7):747-56. doi: 10.1016/S1470-2045(14)70160-3. Epub 2014 Apr 30. PMID 24794243
- [Derived] Hahnen E, Lederer B, Hauke J, Loibl S, Krober S, Schneeweiss A, Denkert C, Fasching PA, Blohmer JU, Jackisch C, Paepke S, Gerber B, Kummel S, Schem C, Neidhardt G, Huober J, Rhiem K, Costa S, Altmuller J, Hanusch C, Thiele H, Muller V, Nurnberg P, Karn T, Nekljudova V, Untch M, von Minckwitz G, Schmutzler RK. Germline Mutation Status, Pathological Complete Response, and Disease-Free Survival in Triple-Negative Breast Cancer: Secondary Analysis of the GeparSixto Randomized Clinical Trial. JAMA Oncol. 2017 Oct 1;3(10):1378-1385. doi: 10.1001/jamaoncol.2017.1007. PMID 28715532